CLINICAL TRIAL: NCT03474055
Title: A Phase II/III, Multicenter, Open-Label, Randomized Study of Liquid Bovine Rotavirus Pentavalent Vaccine (LBRV-PV) to Evaluate Lot-to-Lot Consistency and to Compare Non-Inferiority With ROTASIIL (Lyophilized BRV-PV) in Healthy Infants in India
Brief Title: Study on Liquid Bovine Rotavirus Pentavalent Vaccine (LBRV-PV) to Evaluate Lot-to-Lot Consistency and to Compare Non-Inferiority With ROTASIIL (Lyophilized BRV-PV) in Healthy Infants in India
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Serum Institute of India Pvt. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ROTA:06
Record Dates: First submitted 2018-02-11; First posted 2018-03-22 (Actual); Last update posted 2018-09-10 (Actual); Status verified 2018-09

CONDITIONS: Rotavirus Gastroenteritis
Keywords: Liquid rotavirus vaccine; LBRV-PV; Gastroenteritis; Diarrhoea
MeSH Terms: conditions — Gastroenteritis; Diarrhea

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- LBRV-PV Lot A (Experimental): The study participants in this arm will receive one of the three liquid rotavirus vaccine lots (LBRV-PV Lot A).
  Interventions: Biological: Liquid Rotavirus Vaccine
- LBRV-PV Lot B (Experimental): The study participants in this arm will receive one of the three liquid rotavirus vaccine lots (LBRV-PV Lot B).
  Interventions: Biological: Liquid Rotavirus Vaccine
- LBRV-PV Lot C (Experimental): The study participants in this arm will receive one of the three liquid rotavirus vaccine lots (LBRV-PV Lot C).
  Interventions: Biological: Liquid Rotavirus Vaccine
- ROTASIIL (Active Comparator): The study participants in this arm will receive ROTASIIL, the licensed lyophilized rotavirus vaccine in India.
  Interventions: Biological: Liquid Rotavirus Vaccine

INTERVENTIONS:
Biological: Liquid Rotavirus Vaccine — Liquid Rotavirus Vaccine and Lyophilized Rotavirus Vaccine
  Other Names: ROTASIIL

SUMMARY:
This study has been designed to compare the liquid formulation of BRV-PV (LBRV-PV) with the lyophilized formulation (ROTASIIL) by testing the vaccine in infants (three doses administered 4 weeks apart, starting at 6-8 weeks of age) in order to demonstrate the non-inferiority in the induction of specific anti-rotavirus IgA antibodies by these vaccines. The study will also evaluate lot-to-lot consistency in the manufacture of LBRV-PV by demonstrating equivalence in the induction of specific anti-rotavirus IgA antibodies across three production lots.

ELIGIBILITY:
Inclusion Criteria:

1. Healthy infants as established by medical history and clinical examination before entering the study.
2. Age: 6-8 weeks at the time of enrollment.
3. Parental ability and willingness to provide informed consent.
4. Parent who intends to remain in the area with the child during the study period.

Exclusion Criteria:

1. Presence of diarrhea or vomiting in the previous 72 hours or on the day of enrollment.
2. Acute disease at the time of enrollment (temporary exclusion)
3. Concurrent participation in another clinical trial at any point throughout the entire time frame for this study
4. History of congenital abdominal disorders, intussusception, or abdominal surgery.
5. Known or suspected impairment of immunological function based on medical history and physical examination.
6. History of any neurologic disorders or seizures.
7. Any medical condition in the parents / infant which, in the judgment of the Investigator, would interfere with or serves as a contraindication to protocol adherence or a participant's parents' ability to give informed consent.

Ages: 6 Weeks to 8 Weeks | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 1500 (Actual)
Dates: Start 2017-10-30 (Actual); Primary Completion 2018-06-25 (Actual); Study Completion 2018-06-25 (Actual)

PRIMARY OUTCOMES:
Immunogenicity of rotavirus vaccine | 28 days post dose 3
  Serum anti- rotavirus IgA antibody concentrations expressed as GMCs for the comparison of LBRV-PV vaccine and ROTASIIL

SECONDARY OUTCOMES:
Immunogenicity Endpoints | 28 days post dose 3
  GMCs of serum anti- rotavirus IgA antibody among the LBRV-PV lots at four weeks after the third vaccination.
Immunogenicity Endpoints | 28 days post dose 3
  Proportion of subjects achieving IgA antibody concentration ≥20 U/ml for the comparison of LBRV-PV and ROTASIIL.

CONTACTS AND LOCATIONS:
Locations (8):
- India (8):
  - Centre for Vaccine Studies, Prasanna School of Public Health, Manipal University, Manipal,, Udupi, Karnataka
  - KEM Hospital Research Centre, Pune, Maharashtra
  - Bharati Vidyapeeth Medical College and Hospital, Pune, Pune, Maharashtra
  - Department of community Medicine, Dr Sushila Nayar School of Public Health, Mahatma Gandhi Institute of Medical Sciences, Sewagram, Wardha, Maharashtra
  - Hakeem Abdul Hameed Centenary Hospital, New Delhi, National Capital Territory of Delhi
  - Sri Ramachandra Medical Centre, Chennai, Chennai, Tamil Nadu
  - Institute of Child Health, Kolkata, Kolkata, West Bengal
  - Post Graduate Institute of Medical Education and Research, Chandigarh, Chandigarh

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Kawade A, Babji S, Kamath V, Raut A, Kumar CM, Kundu R, Venkatramanan P, Lalwani SK, Bavdekar A, Juvekar S, Dayma G, Patil R, Kulkarni M, Hegde A, Nayak D, Garg BS, Gupta S, Jategaonkar S, Bedi N, Maliye C, Ganguly N, Uttam KG, Niyogi P, Palkar S, Hanumante N, Goyal N, Arya A, Aslam M, Parulekar V, Dharmadhikari A, Gaikwad D, Zade J, Desai S, Kang G, Kulkarni PS. Immunogenicity and lot-to-lot consistency of a ready to use liquid bovine-human reassortant pentavalent rotavirus vaccine (ROTASIIL - Liquid) in Indian infants. Vaccine. 2019 May 1;37(19):2554-2560. doi: 10.1016/j.vaccine.2019.03.067. Epub 2019 Apr 4. PMID 30955982